CLINICAL TRIAL: NCT02872909
Title: A Randomized Assessor-blinded Comparison of Low Irradiance and Conventional Irradiance Photodynamic Therapy (PDT) for Superficial Non-melanoma Skin Cancer
Brief Title: Randomized Comparison of Low and Conventional Irradiance PDT for Skin Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sally Ibbotson (Other)
Responsible Party: Sponsor-Investigator, Sally Ibbotson, Dr Sally H Ibbotson, University of Dundee
Organization: University of Dundee (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011DS04
Record Dates: First submitted 2016-08-05; First posted 2016-08-19 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- low irradiance LED PDT (Active Comparator): Ambulight LED portable PDT treatment
  Interventions: Device: Ambulight (Ambicare Health)
- conventional higher irradiance LED (Active Comparator): Conventional LED hospital based standard PDT treatment
  Interventions: Device: Ambulight (Ambicare Health)

INTERVENTIONS:
Device: Ambulight (Ambicare Health) — battery-operated low irradiance red light LED ("skin cancer plaster")

SUMMARY:
This study aims to examine whether the pain of topical photodynamic therapy (PDT) is significantly different when using low irradiance ambulatory light emitting diode (LED) devices compared with conventional higher irradiance hospital based LED light sources when used for superficial non-melanoma skin cancer. The investigators are also investigating the phototoxicity and efficacy of each regime in this randomized assessor-blinded clinical trial.

DETAILED DESCRIPTION:
A randomized assessor-blinded comparative study of low irradiance ambulatory LED devices with conventional hospital-based LED devices for superficial non-melanoma skin cancer. Preliminary observations suggest that low irradiance LEDs cause less pain but are as effective, so the investigators are examining this in a clinical trial of patients with lesions </= 2cm diameter of non-melanoma skin cancer (Bowen's disease and superficial basal cell carcinoma). Patients with these conditions referred to the PDT clinic will be invited to participate and if they are eligible and consent to treatment then they will be prospectively randomized to either ambulatory PDT or conventional PDT. Pain and phototoxicity scores will be recorded and clinical efficacy will be assessed up to one year after the last treatment. Computer-generated block randomization will be performed and at 90% power to detect as significant at the 5% level a mean difference in pain score of 2 in one group compared with 4 in the other, 36 patients will be needed, and as the participants will often be elderly and frail the investigators will aim for a safety margin of recruiting 50 participants to account for drop-outs. Participants will receive two treatments of either arm at a one week interval and will be assessed clinically at three months and if residual disease remains then the two treatments a week apart are repeated. Pain assessed using a visual analogue scale (VAS) score and phototoxicity on a semi-quantitative scale are recorded at 7 days when the participant returns for their second treatment. Follow up for clinical assessment is at 6 months and one year after treatment. Participants also give their opinion of treatment at one year follow up. Assessors of adverse effects and efficacy will be blinded. Data recording and analysis will be undertaken by the study statistician Dr Robert Dawe and analysis will be on an intention to treat basis using appropriate statistical tests comparing the pre-planned outcome measures, with pain as primary outcome and outcome, efficacy and patient satisfaction as secondary outcomes

ELIGIBILITY:
Inclusion Criteria:

* Bowen's disease or superficial basal cell carcinoma referred for PDT and lesion not greater than 2.4cm diameter

Exclusion Criteria:

* Unable to give consent, >2cm diameter, lesions on highly curved surfaces where ambulatory device would not adhere

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sally H Ibbotson, MD, Principal Investigator — University of Dundee

IPD SHARING:
Plan to Share IPD: Yes
peer reviewed publications and presentations at international and national meetings
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: presenting study data at British Association of Dermatologists annual meeting Edinburgh 5.7.18 and abstract will be published in Br J Dermatol and full publication will follow
Access Criteria: via presentation and publication in peer-reviewed journal

REFERENCES:
- [Background] Attili SK, Lesar A, McNeill A, Camacho-Lopez M, Moseley H, Ibbotson S, Samuel ID, Ferguson J. An open pilot study of ambulatory photodynamic therapy using a wearable low-irradiance organic light-emitting diode light source in the treatment of nonmelanoma skin cancer. Br J Dermatol. 2009 Jul;161(1):170-3. doi: 10.1111/j.1365-2133.2009.09096.x. Epub 2009 Mar 19. PMID 19302071
- [Background] Moseley H, Allen JW, Ibbotson S, Lesar A, McNeill A, Camacho-Lopez MA, Samuel ID, Sibbett W, Ferguson J. Ambulatory photodynamic therapy: a new concept in delivering photodynamic therapy. Br J Dermatol. 2006 Apr;154(4):747-50. doi: 10.1111/j.1365-2133.2006.07145.x. PMID 16536822
- [Background] Ibbotson SH. Irradiance is an important determinant of pain experienced during topical photodynamic therapy. J Am Acad Dermatol. 2011 Jul;65(1):201-2. doi: 10.1016/j.jaad.2010.11.060. No abstract available. PMID 21679812
- [Background] Ibbotson SH, Ferguson J. Ambulatory photodynamic therapy using low irradiance inorganic light-emitting diodes for the treatment of non-melanoma skin cancer: an open study. Photodermatol Photoimmunol Photomed. 2012 Oct;28(5):235-9. doi: 10.1111/j.1600-0781.2012.00681.x. PMID 22971187

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
Started | 32 | 18
Completed | 32 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED | Total
Number analyzed (Participants) | 32 | 18 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 12
  >=65 years | 22 | 16 | 38
Age, Continuous [Median (Full Range); unit: years] | 75 [41 to 87] | 71 [59 to 83] | 71 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 12 | 35
  Male | 9 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Technical failure with ambulatory devices in first two participants meant that no data could be evaluated for these first two recruited subjects
  participants
    United Kingdom | 34 | 18 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pain on VAS Score
Description: assess on visual analogue scale (VAS) score of 0 - 10cm, with 0 representing no pain experienced through to 10 representing the worst pain imaginable. The participant marks across a 0-10cm unmarked line where their level of pain experience is and this is measured eg. 2cm if experiencing mild pain or 8.5cm which would represent severe pain
Time Frame: one week after treatment
Population: The ambulatory devices suffered technical failure in the first two participants so no data were available for these subjects. Data were available for 32 participants treated with ambulatory PDT and 18 treated with conventional PDT
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
Number analyzed (Participants) | 32 | 18
score on a scale | 2.95 [0.5 to 4.8] | 1.25 [0.7 to 2.8]
Statistical Analysis 1: Comparison: Low Irradiance LED PDT vs Conventional Higher Irradiance LED; Sample size requirement estimation - Preliminary data showed pain scores of 1.25 with ambulatory PDT (n=12) and 5.26 (SD 2.38) for conventional PDT (n=50). Estimated that for 85% power to detect as significant at 5% level a difference in mean pain score in one group of 2cm compared with 4 cm in the other group, assuming two-sided testing, a minimum of 45 subjects needed. We aimed for 50 subjects, with an allocation ratio of 2 (twice as many randomised to ambulatory PDT as conventional PDT); Test type: Superiority; p < 0.05, t-test, 2 sided — calculated as <0.05 for 85% power; Analysed on log transformed data; Mean Difference (Final Values) = 1.37, 95% CI 2-sided [0.71 to 2.54]

2. Secondary Outcome: Phototoxicity
Description: erythema, oedema, blistering, crusting, ulceration on semi-quantitative scale. Erythema is graded as 0 = absent, 1 = mild, 2 = moderate or 3 = severe erythema as assessed by naked eye examination. Oedema is graded as 0 = absent or 1 = present. Likewise crusting or ulceration are each graded as 0 = absent and 1 = present by naked eye examination. Data will be presented and analysed separately ie. erythema data will be presented and then separately whether oedema, crusting or ulceration are present or absent.
  ie. reporting may appear as example: erythema score 3 of range of 0-3 options; oedema score 1 (binary option of 0 or 1); crusting score 0 (binary option of 0 or 1); ulceration score 0 (binary option of 0 or 1)
Time Frame: one week after treatment
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
Number analyzed (Participants) | 32 | 18
score on a scale | 2 [0 to 3] | 1 [0 to 3]

3. Secondary Outcome: Clinical Clearance of Lesion
Description: clinical assessment by study dermatologist to determine by inspection and palpation whether the lesion is clear, partially clear or not clear - assessed at 3, 6 and 12 months after treatment, with 12 months as the final study outcome endpoint analysed
Time Frame: 12 months after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
Number analyzed (Participants) | 32 | 18
Participants | 27 | 14

4. Secondary Outcome: Patient Satisfaction
Description: brief patient questionnaire to evaluate their opinion of the treatment they received. This is assessed as A.efficacy of treatment - 1 = not effective NR; 2 = partIally effective PR; 3 = completely effective CR; B.Side effects of treatment eg. pain and inflammation - 1 = severe; 2 = moderate; 3 = mild; 4 = none/minimal. C.Practicalities of treatment eg. ease of use, travel, time, inconvenience - 1 = very disruptive and difficult; 2 = moderately disruptive and difficult; 3 = minimally disruptive and difficult. The scores of A, B and C will be added to give an overall score with range of overall minimum score option 3 and maximum 10.
  Patients will also separately be asked to give overall evaluation on a VAS scale of 0 = treatment very poor and would not have again through to 10 = treatment excellent and I would have again - with a continuous line option from 0 - 10 to mark across, providing a separate score with range options 0 to 10
Time Frame: one year after treatment - last visit
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
Number analyzed (Participants) | 32 | 18
score on a scale | 10 [5.5 to 10] | 10 [8 to 10]
Statistical Analysis 1: Comparison: Low Irradiance LED PDT vs Conventional Higher Irradiance LED; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up to 1 year follow up visit for each participant
Arm/Group | Low Irradiance LED PDT | Conventional Higher Irradiance LED
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/18
Other Adverse Events (participants affected / at risk) | 0/32 | 0/18

LIMITATIONS AND CAVEATS:
Nil of note

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT02872909/Prot_SAP_000.pdf